CLINICAL TRIAL: NCT00406107
Title: Open Label Macugen for the Treatment of Macular Edema Secondary to Branch Retinal Vein Occlusion
Brief Title: Evaluation of Macugen Treatment of Macular Edema Due to Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Palmetto Retina Center, LLC (Other)
Collaborators: Pfizer (Industry); Eyetech Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, John A. Wells, III, M.D., Principal Investigator, Palmetto Retina Center, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRC-001; Pfizer Reference # 20050548
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: branch retinal vein occlusion; macular edema; pegaptanib sodium; vascular endothelial growth factor
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegaptanib Sodium 0.3mg (Macugen) (Active Comparator): Intravitreous injections of Macugen 0.3mg given at baseline, week 6 and week 12 with subsequent injections at six weekly intervals at the discretion of the investigator until week 54.
  Interventions: Drug: pegaptanib sodium (Macugen)
- Pegaptanib Sodium 1 mg (Macugen) (Active Comparator): Intravitreous injections of Macugen 1.0mg given at baseline, week 6 and week 12 with subsequent injections at six weekly intervals at the discretion of the investigator until week 54.
  Interventions: Drug: pegaptanib sodium (Macugen)

INTERVENTIONS:
Drug: pegaptanib sodium (Macugen) — Subjects were randomized 3:1 to intravitreous injections of pegaptanib 0.3mg or 1mg at baseline and at weeks 6 and 12 with subsequent injections at 6-week intervals at investigator discretion until week 48.
  Other Names: Macugen

SUMMARY:
The purpose of this study is to evaluate the effect of intravitreal injections of Macugen every 6 weeks for the treatment of macular edema secondary to branch retinal vein occlusion (BRVO). We hypothesize that macular edema secondary to BRVO is mediated by VEGF 165 and that chronic suppression of VEGF 165 will successfully treat BRVO related macular edema.

DETAILED DESCRIPTION:
Retinal venous occlusive disease, which includes central retinal vein occlusion (CRVO) and branch retinal vein occlusion (BRVO), is second only to diabetic retinopathy as a cause of vision loss due to retinal disease. The main cause of vision loss in all of these disorders is the development of macular edema. Current clinical practice based on randomized controlled clinical trials (ETDRS, BVOS) employs laser photocoagulation, either in a focal or grid pattern, to treat macular edema associated with diabetic retinopathy and branch retinal vein occlusion. Unfortunately, laser photocoagulation is ineffective in central retinal vein occlusion (CRVO), and no proven therapy exists for CRVO.

The pathogenesis of macular edema in retinal vascular diseases is generally accepted to be increased levels of vascular endothelial growth factor (VEGF) due to ischemic or other stimuli. VEGF is known to be one of the most potent stimulators of vascular leakage in humans. Therefore, it seems sensible to study inhibition of VEGF to reduce vascular leakage, reduce macular edema, and improve vision in these retinal vascular disorders.

Phase 2 randomized, controlled clinical trials of Macugen in diabetic macular edema and in macular edema associated with CRVO have been conducted. In the diabetes trial, patients treated with Macugen had improved vision, reduced macular edema as measured by optical coherence tomography (OCT), and reduced need for laser treatment compared to patients treated with sham injections. In the CRVO trial, patients treated with Macugen 1 mg every 6 weeks for 24 weeks had improved vision and reduced macular edema at week 30 compared to sham. This is the first randomized trial of treatment for CRVO to show a benefit over control. Based on these positive findings, we plan to study Macugen treatment of macular edema due to BRVO.

ELIGIBILITY:
Inclusion Criteria:

* Macular edema secondary to BRVO involving the foveal center in male or female patients at least 18 years of age
* Duration of BRVO macular edema less than 6 months prior to baseline visit
* Best corrected ETDRS visual acuity 20/40-20/320 (Snellen equivalent) using the 4 meters testing method.
* Central foveal thickness greater than or equal to 250 microns using the OCT-3
* Less than 25% of foveal capillary ring disruption
* Less than 2 disc areas of capillary non-perfusion within 1000 microns of the foveal center
* Absence of hemorrhage or lipid in the foveal center
* Investigator comfortable deferring macular laser for 18 weeks from baseline and intravitreous steroid for 36 weeks from baseline

Exclusion Criteria:

* Ocular conditions other than BRVO related macular edema such as significant cataract, diabetic retinopathy, AMD, glaucoma, uveitis, epiretinal membrane, vitreomacular traction or tumor.
* Intraocular surgery within past 3 months
* Significant enlargement of foveal avascular zone(>25% disruption of capillary ring) or greater than 2 disc areas of nonperfusion within 1000 microns of foveal center.
* Likelihood of evidence driven indication for peripheral photocoagulation in the next 6 months.
* Patients who have shown evidence of spontaneous improvement within the preceding 3 months, as determined by an improvement of >15 letters of vision or thinning of the Center Point on OCT of >20% from baseline determination
* Prior grid laser within 4 months of baseline or more than one prior grid laser treatment.
* No prior intravitreous or periocular steroid injections in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Wells, III, MD, Principal Investigator — Palmetto Retina Center, LLC
Locations (3):
- United States (3):
  - Jules Stein Eye Institute, Los Angeles, California
  - Cumberland Valley Retina Center, Hagerstown, Maryland
  - Palmetto Retina Center, West Columbia, South Carolina

REFERENCES:
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Argon laser photocoagulation for macular edema in branch vein occlusion. The Branch Vein Occlusion Study Group. Am J Ophthalmol. 1984 Sep 15;98(3):271-82. doi: 10.1016/0002-9394(84)90316-7. PMID 6383055
- [Background] Evaluation of grid pattern photocoagulation for macular edema in central vein occlusion. The Central Vein Occlusion Study Group M report. Ophthalmology. 1995 Oct;102(10):1425-33. doi: 10.1016/s0161-6420(95)30849-4. PMID 9097788
- [Background] Cunningham ET Jr, Adamis AP, Altaweel M, Aiello LP, Bressler NM, D'Amico DJ, Goldbaum M, Guyer DR, Katz B, Patel M, Schwartz SD; Macugen Diabetic Retinopathy Study Group. A phase II randomized double-masked trial of pegaptanib, an anti-vascular endothelial growth factor aptamer, for diabetic macular edema. Ophthalmology. 2005 Oct;112(10):1747-57. doi: 10.1016/j.ophtha.2005.06.007. PMID 16154196
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Funatsu H, Yamashita H, Ikeda T, Nakanishi Y, Kitano S, Hori S. Angiotensin II and vascular endothelial growth factor in the vitreous fluid of patients with diabetic macular edema and other retinal disorders. Am J Ophthalmol. 2002 Apr;133(4):537-43. doi: 10.1016/s0002-9394(02)01323-5. PMID 11931788

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegaptanib Sodium 0.3mg (Macugen) | Pegaptanib Sodium 1 mg (Macugen)
Started | 15 | 5
Completed | 14 | 4
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pegaptanib Sodium 1 mg (Macugen): Intravitreous injections of Macugen 1.0 mg given at baseline, week 6 and week 12 with subsequent injections at six weekly intervals at the discretion of the investigator until week 54.
- Total: Total of all reporting groups
Arm/Group | Pegaptanib Sodium 0.3mg (Macugen) | Pegaptanib Sodium 1 mg (Macugen) | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 12 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (8.2) | 77 (8.7) | 73.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in ETDRS Best Corrected Visual Acuity From Baseline at 54 Weeks
Time Frame: 54 Weeks
Measure: Mean (Standard Deviation); unit: ETDRS letters
Groups:
- All Study Participants: Outcome measures were assessed without regard to dosage of pegaptanib received
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
ETDRS letters | 14 (13)

2. Secondary Outcome: Standardized Change From Baseline in Macular Thickening Measured by OCT3 Using the Central Point of the Central Subfield
Time Frame: 54 Weeks
Population: Fifteen patients were enrolled in the pegaptanib 0.3 mg dose group and 5 patients were enrolled in the 1.0 mg dose group.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
microns | -205 (195)

3. Secondary Outcome: Safety Parameters
Description: Safety endpoints incuded all investigator reported ocular and systemic adverse events. All events were graded as mild moderate or severe and assessed as related or unrelated to the injection procedure and the study drug.
Time Frame: 54 Weeks
Measure: Number; unit: percentage of participants
Groups:
- Pegaptanib Sodium 0.3mg (Macugen): Patients experiencing an ocular adverse event, in this case a retinal detachment
Arm/Group | Pegaptanib Sodium 0.3mg (Macugen) | Pegaptanib Sodium 1 mg (Macugen)
Number analyzed (Participants) | 15 | 5
percentage of participants | 6.67 | 0

4. Secondary Outcome: Change in Central Subfield Thickness on OCT From Baseline to Week 54
Time Frame: 54 Weeks
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
microns | -201 (153)

5. Secondary Outcome: Change in Macular Volume on OCT From Baseline to Week 54
Time Frame: 54 Weeks
Measure: Mean (Standard Deviation); unit: mm cubed
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
mm cubed | -2.2 (1.6)

ADVERSE EVENTS:
Arm/Group | Pegaptanib Sodium 0.3mg (Macugen) | Pegaptanib Sodium 1 mg (Macugen)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 1/15 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegaptanib Sodium 0.3mg (Macugen) (N=15) | Pegaptanib Sodium 1 mg (Macugen) (N=5)
retinal detachment (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No